CLINICAL TRIAL: NCT06169813
Title: Evaluating Smoking Cessation and Harm Reduction Approaches Among People Living With HIV/AIDS in South Africa
Brief Title: E-cigarette Harm Reduction Among PLWHA in South Africa
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-00868
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking | interventions — Nicotine Replacement Therapy; Electronic Nicotine Delivery Systems; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Quit-Line Referral) (Active Comparator): Participants will receive referral to the existing South African Quitline. Participants will receive information to contact the Quitline if participants so choose, in addition to ecological momentary assessment (EMA) texting orientation.
  Interventions: Behavioral: Counseling
- Nicotine Replacement Therapy (NRT) (Experimental): In addition to phone counseling + ecological momentary intervention (EMI) texting, participants will receive combination NRT (daily patches and lozenges).
  Interventions: Other: Nicotine Replacement Therapy (NRT); Behavioral: Counseling
- Electronic Cigarette (EC) (Experimental): In conjunction with phone counseling + EMI texting, participants will receive the VUSE "Solo" EC.
  Interventions: Other: E-Cigarette (EC); Behavioral: Counseling

INTERVENTIONS:
Other: Nicotine Replacement Therapy (NRT) — NRT (daily patches and lozenges). NRT strength will be according to the established dosing guidelines for tobacco treatment. NRT is the standard of care in tobacco treatment and helped reduce CPD in prior trials
  Arms: Nicotine Replacement Therapy (NRT)
Other: E-Cigarette (EC) — EC with single-use pods. Nicotine - 48 mg/ ml (4.8% nicotine) concentration.
  Other Names: Vuse Solo EC
  Arms: Electronic Cigarette (EC)
Behavioral: Counseling — Each participant will receive up to 5-motivational counseling sessions. The first session will also include orientation of EMA/EMI texting.

SUMMARY:
The purpose of this pilot randomized controlled trial study aims to address the unmet need for feasible and efficacious strategies for reducing combustible cigarette (CC) use among people living with HIV/AIDS (PLWHA) in South Africa, which has the potential to significantly improve the health and long-term survival of PLWHA CC smokers. Using the proposed intervention, based on the Information-Motivation-Behavioral Skills (IMB), and a simultaneous embedded mixed methods approach, the investigators will evaluate a telehealth program targeting CC harm reduction, comparing E-cigarettes (EC) to nicotine replacement therapy (NRT) that is enhanced by integrating ecological momentary intervention (EMI) texting. As such, this proposal will significantly build research capacity in South Africa to conduct telehealth tobacco treatment interventions using innovative EMI approaches enhancing participants' engagement, as well as state-of-the art evaluation approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adult PLWHA CC smokers;
* Speaks Afrikaans, or Xhosa, or English;
* reports daily CC smoking (≥ 5 CPD);
* Owns any type of mobile phone;
* interested in reducing CC smoking but not necessarily trying to quit;
* Receives HIV/AIDS care in one of the eight selected clinics follow-up rates.

Exclusion Criteria:

* are pregnant or breastfeeding;
* unable to provide consent;
* used tobacco products other than CC in the past 2 weeks (e.g., EC, cigarillo);
* currently engaged in an attempt to quit CC smoking;
* current major depressive or manic episode, current psychotic disorder, past-year suicide attempt, or current suicidal ideation with plan or intent. plan or intent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Up to Month 6
  Defined as the total number of participants recruited divided by the maximum number of recruiting sites, then divided by the total number of months that the trial recruited for.
Percent of Patients who Enroll in Counseling | Up to Month 6
  Defined as the percentage of participants who start the intervention counseling sessions.
Follow-Up Rate at 3 Months | Month 3
  Defined as the percent of participants who completed the 3-month follow-up.
Follow-Up Rate at 6 Months | Month 6
  Defined as the percent of participants who completed the 6-month follow-up.
Client Satisfaction Questionnaire (CSQ-8) Score | Week 8
  8-item assessment of satisfaction with the intervention. The total score is the sum of responses and ranges from 8 to 32, with higher numbers indicating greater satisfaction.
Client Satisfaction Questionnaire (CSQ-8) Score | Month 3
  8-item assessment of satisfaction with the intervention. The total score is the sum of responses and ranges from 8 to 32, with higher numbers indicating greater satisfaction.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve 7-Day Point Prevalence Abstinence. | Month 3
  Abstinence will be verified by exhaled carbon monoxide and defined as no combustible cigarette use in the last 7 days.
Percentage of Participants who achieve 50% Reduction in Cigarettes Per Day (CPD), compared with Baseline | Up to Month 6
  CPD will be self-reported.
Change in American Thoracic Society Questionnaire Score | Baseline, Month 6
  Change in American Thoracic Questionnaire Score from Baseline to Week 12 8-item questionnaire assessing general thoracic pain. Items are rated on a Likert scale from 1 (never) to 5 (every day). The total score is the sum of responses and ranges from 8-40; higher scores indicate more severe impact of general thoracic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Omar El-Shahawy, Principal Investigator — NYU Langone Health
Locations (1):
- South African Medical Research Council (SAMRC), Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request or for individual participant data meta-analysis beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data or the researchers who provide a methodologically sound proposal execute a data use agreement with NYU Langone Health. Requests may be directed to: Omar.ElShahawy@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data or the researchers who provide a methodologically sound proposal will be granted access upon reasonable request or for individual participant data meta-analysis. Requests should be directed to Omar.ElShahawy@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT06169813/ICF_000.pdf